CLINICAL TRIAL: NCT03269435
Title: A Randomized Trial of Greater Occipital Nerve Block With Bupivacaine Versus Intravenous Metoclopramide for Acute Migraine
Brief Title: Greater Occipital Nerve Block Versus Metoclopramide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-8249
Record Dates: First submitted 2017-08-18; First posted 2017-08-31 (Actual); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Bupivacaine; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double dummy design with IV placebo and placebo nerve block
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Greater Occipital Nerve Block (Experimental): Bilateral greater occipital nerve block with bupivacaine 0.5%
  + Normal saline IV
  Interventions: Procedure: Greater occipital nerve block with bupivacaine
- Metoclopramide (Active Comparator): Metoclopramide 10mg IV
  + Bilateral greater occipital nerve block with normal saline
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Procedure: Greater occipital nerve block with bupivacaine — This is a type of peripheral nerve block. 3cc of 0.5% bupivacaine will be injected adjacent to the greater occipital nerve block blaterally
  Arms: Greater Occipital Nerve Block
Drug: Metoclopramide — Metoclopramide 10mg IV will be administered over 15 minutes
  Arms: Metoclopramide

SUMMARY:
We are comparing a type of nerve block called greater occipital nerve block versus standard therapy among patients who present to an emergency department for acute migraine. This is a randomized, double-blind, double dummy study. The greater occipital nerve block will be performed bilaterally with bupivacaine 0.5%. Standard therapy is metoclopramide 10mg IV.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients are adults who present with an acute moderate or severe headache meeting migraine headache criteria, as defined by the International Classification of Headache Disorders-3β (1.1, migraine without aura). Patients who meet criteria for Probable Migraine without Aura (1.5.1) will also be included, provided they have had at least one similar attack previously.

Exclusion Criteria:

Patients will be excluded if informed consent cannot be obtained, if there is concern for a secondary cause of headache, if the maximum documented temperature is greater than 100.3 degrees, for a new objective neurologic abnormality, skull defect, suspected infection overlying injection site, known bleeding disorder, ongoing use of anti-platelet agents including P2Y12 platelet inhibitors (clopidogrel, prasugrel, ticagrelor), heparins, warfarin, or 10a inhibitors (rivaroxaban, apixaban, edoxaban, fondaparinux), prior treatment with a greater occipital nerve block, allergy to the investigational medications, pheochromocytoma, seizure disorder, Parkinson's disease, use of MAO inhibitors, and use of anti-rejection transplant medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-described
Enrollment: 99 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Greater Occipital Nerve Block: Bilateral greater occipital nerve block with bupivacaine 0.5%
  + Normal saline IV
  Greater occipital nerve block with bupivacaine: This is a type of peripheral nerve block. 3cc of 0.5% bupivacaine will be injected adjacent to the greater occipital nerve block blaterally
- Metoclopramide: Metoclopramide 10mg IV
  + Bilateral greater occipital nerve block with normal saline
  Metoclopramide: Metoclopramide 10mg IV will be administered over 15 minutes
Period: Overall Study
Arm/Group | Greater Occipital Nerve Block | Metoclopramide
Started | 51 | 48
Completed | 51 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Greater Occipital Nerve Block | Metoclopramide | Total
Number analyzed (Participants) | 51 | 48 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (11) | 38 (11) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 34 | 78
  Male | 7 | 14 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 48 | 99
Baseline pain intensity [Count of Participants; unit: Participants]
  Severe pain | 38 | 35 | 73
  Moderate pain | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: 0-10 Pain Score
Description: Pain score assessed at baseline and one hour. 0= no pain, 10 = worst imaginable. This outcome is the change in pain between baseline and one hour
Time Frame: one hour
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Greater Occipital Nerve Block | Metoclopramide
Number analyzed (Participants) | 51 | 48
units on a scale | 5.0 [4.1 to 5.8] | 6.1 [5.2 to 6.9]

2. Secondary Outcome: Sustained Headache Relief
Description: Headache level = mild or none. Achieved in emergency department and maintained for 48 hours without rescue medication
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve Block | Metoclopramide
Number analyzed (Participants) | 51 | 47
Participants | 11 | 18

3. Secondary Outcome: Sustained Headache Freedom
Description: Headache = none, achieved in emergency department and maintained for 48 hours
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve Block | Metoclopramide
Number analyzed (Participants) | 51 | 48
Participants | 3 | 7

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Greater Occipital Nerve Block | Metoclopramide
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 16/51 | 18/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Greater Occipital Nerve Block (N=51) | Metoclopramide (N=48)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
drowsiness (Nervous system disorders) | 0 (0) | 3 (3)
headache (Nervous system disorders) | 3 (3) | 2 (2)
head numbness (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Injection site reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Gastrointestinal symptoms (Gastrointestinal disorders) | 2 (2) | 0 (0)
Various (Investigations) | 1 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03269435/Prot_SAP_000.pdf